CLINICAL TRIAL: NCT03269565
Title: An International Multicenter Open-label Randomized Trial of the Efficacy, Pharmacokinetics, Safety, and Immunogenicity of BCD-100 (JSC BIOCAD, Russia) as Monotherapy in Patients With Unresectable/Metastatic Melanoma.
Brief Title: International Trial of the Efficacy and Safety of BCD-100 in Patients With Melanoma
Acronym: MIRACULUM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-100-2
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): BCD-100 1 mg/kg Q2W;
  Interventions: Biological: BCD-100
- Arm 2 (Experimental): BCD-100 3 mg/kg Q3W.
  Interventions: Biological: BCD-100

INTERVENTIONS:
Biological: BCD-100 — Anti-PD-1 monoclonal antibody

SUMMARY:
An International Multicenter Open-label Randomized Trial of the Efficacy, Pharmacokinetics, Safety, and Immunogenicity of BCD-100 (JSC BIOCAD, Russia) as Monotherapy in Patients with Unresectable/Metastatic Melanoma.

DETAILED DESCRIPTION:
This trial has been designed as an international multicenter open-label Phase II trial.

The trial aims to investigate the efficacy, pharmacokinetics, safety, and immunogenicity of two dosage regimens of BCD-100 (JSC BIOCAD, Russia) as monotherapy in patients with unresectable/metastatic melanoma.

According to the design, the trial will include two arms of patients. Each of the trial arms will receive repeated doses of the test drug as monotherapy; BCD-100 will be administered using one of the following dosage regimens established in a Phase I trial:

* Monotherapy, BCD-100 1 mg/kg Q2W (IV infusion over 60 minutes; if a 60-minute infusion is tolerated well, all following doses can be administered over 30 minutes);
* Monotherapy, BCD-100 3 mg/kg Q3W (IV infusion over 60 minutes; if a 60-minute infusion is tolerated well, all following doses can be administered over 30 minutes).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form and the subject's ability to follow the Protocol requirements;
2. Age: 18 years and older at the signing of the informed consent;
3. Histologically verified (documented) unresectable/metastatic melanoma;
4. Newly diagnosed advanced/metastatic melanoma or progressive disease during (or after) systemic chemotherapy ;
5. Available tissue blocks for histological examination or patient's agreement to give biopsy specimens for PD-L1 expression status ;
6. ECOG performance status of 0 or 1;
7. LDH less than or equal to 2×upper limit of normal;
8. At least one RESICT 1.1-defined measurable target lesion confirmed by an independent review;
9. All prior treatment-related toxicities/surgery-related adverse events must be less than or equal to Grade 2 according to CTCAE 4.03, except for chronic/permanent damage caused by an AE that does not affect the safety profile of the investigational therapy (e.g., alopecia);
10. Adequate organ system function ;
11. Life expectancy of at least 12 weeks from the screening.
12. Patients with reproductive potential must agree to practice acceptable methods of birth control throughout the entire trial period, starting from signing the informed consent and up to 12 weeks after the last dose of BCD-100.

Exclusion Criteria:

1. Evidence of severe or concomitant diseases/life-threatening complications of the main condition (e.g., massive pleural, pericardial, or peritoneal effusion that requires medical intervention , pulmonary lymphangitis) at the signing of the informed consent;
2. Subjects with progressive/symptomatic brain metastases (e.g., brain edema, spinal cord compression) or brain metastases that need therapy with corticosteroids and/or anticonvulsants ;
3. Any concomitant disease observed at the screening that increases the risk of adverse events during the investigational therapy:

   * Grade III-IV stable angina, unstable angina, or a history of myocardial infarction within 6 months prior to signing the informed consent;
   * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system;
   * Severe, resistant hypertension;
   * History of atopic asthma, angioedema;
   * Moderate to severe respiratory failure, Grade 3 to 4 chronic obstructive pulmonary disease;
   * Any other concomitant condition (e.g., metabolism, blood, hepatic, renal, pulmonary, neurological, endocrine, cardiac, infectious, or gastrointestinal disorder) that constitutes an unacceptable risk to the patient's health during the investigational therapy;
4. Systemic autoimmune diseases (including but not limited to SLE, Crohn's disease, ulcerative colitis, systemic scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, etc.) ;
5. Endocrine disorders that cannot be adequately controlled by hormone replacement therapy without any dose modification within 28 days prior to the start of the investigational therapy;
6. Patients who need therapy with corticosteroids or other immunosuppressants;
7. Blood disorders :

   * Neutrophils <1.5×109/L;
   * Platelets <100×109/L;
   * Hb <90 g/L;
8. Impaired renal function: creatinine ≥1.5×ULN;
9. Impaired liver function :

   * Bilirubin ≥1.5×ULN (≤50 μmol/L for patients with Gilbert's syndrome);
   * AST/ALT ≥2.5×ULN (5×ULN for patients with liver metastases);
   * ALP ≥5×ULN;
10. LDH >2×ULN;
11. Anti-cancer therapy (surgery, chemotherapy) within 28 days prior to the first dose of the investigational product; radiotherapy within 14 days prior to the first dose of the investigational product;
12. Prior treatment with anti-CTLA4 and/or anti-PD-1/PD-L1/PD-L2 agents;
13. Prior targeted therapy ;
14. Patients who have received more than two lines of systemic chemotherapy for unresectable or metastatic melanoma;
15. Concomitant cancer (except for cervical carcinoma in situ after radical surgery or basal cell/squamous cell carcinoma after radical surgery);
16. Any condition that prevents a patient from following the Protocol procedures (dementia, neurological or mental disorders, drug/alcohol abuse, etc.) ;
17. Simultaneous participation in other clinical trials , participation in other clinical trials within 30 days prior to the first dose of the investigational product;
18. Acute infection or the acute phase of chronic infection within 28 days prior the first dose of the investigational product;
19. Active HBV/HCV/HIV infection, active syphilis ;
20. Patients unable to receive an IV infusion of BCD-100;
21. Patients unable to receive an IV contrast agent;
22. Hypersensitivity to any of the components of BCD-100;
23. History of hypersensitivity to any therapeutic monoclonal antibody;
24. Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  Overall response rate (partial response+complete response rates) assessed according to irRECIST in an mITT population during BCD-100 therapy

SECONDARY OUTCOMES:
One-year progression-free survival rate ; | 1 year
  One-year progression-free survival rate during BCD-100 therapy;
Percentage of patients with severe immune-related AEs | 1 year
  Percentage of patients with severe immune-related AEs (CTCAE 4.03 Grade 3 or greater);

CONTACTS AND LOCATIONS:
Overall Officials: Yulia N Linkova, MD, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (9):
- Russia (9):
  - State Budgetary Institution of Healthcare of the Arkhangelsk Region "Arkhangelsk Regional Clinical Oncology Dispensary" (SBHI AR ARCOD), Arkhangelsk
  - "N.N. Blokhin Russian Cancer Research Center", Moscow
  - State Budgetary Healthcare Institution "Moscow Clinical Scientific Center funded by Moscow Health Department" (SBHI MCSC MHD), Moscow
  - "Pavlov First Saint Petersburg State Medical University", Saint Petersburg
  - "Saint Petersburg Clinical Research and Practice Center for Specialized Medical Care (Oncology)", Saint Petersburg
  - Federal State Budgetary Institution "N.N. Petrov Research Institute of Oncology" of the Ministry of Healthcare of the Russian Federation (FSBI N.N. Petrov RIO (Chemotherapy Department with Innovative Technologies), Saint Petersburg
  - Federal State Budgetary Institution "N.N. Petrov Research Institute of Oncology" of the Ministry of Healthcare of the Russian Federation, Research Department of the Innovative Methods of Therapeutic Oncology and Rehabilitation (FSBI N.N. Petrov RIO of the, Saint Petersburg
  - LLC BioEk, Saint Petersburg
  - State Budgetary Institution of Healthcare "Clinical Oncology Dispensary of Chelyabinsk Region" (SBIH CODCR), Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demidov L, Kharkevich G, Petenko N, Moiseenko V, Protsenko S, Semiglazova T, Zimina A, Kovalenko N, Fadeeva N, Kirtbaya D, Belogortsev I, Tantsyrev D, Odintsova S, Nesterova A, Vorontsova K, Makarycheva Y, Linkova Y, Zinkina-Orikhan A, Siliutina A, Sorokina I, Liaptseva D, Chistyakov V, Lutsky A. A phase III study to access the safety and efficacy of prolgolimab 250 mg fixed dose administered every 3 weeks versus prolgolimab 1 mg/kg every 2 weeks in patients with metastatic melanoma (FLAT). Front Oncol. 2024 Sep 4;14:1385685. doi: 10.3389/fonc.2024.1385685. eCollection 2024. PMID 39296979
- [Derived] Tjulandin S, Demidov L, Moiseyenko V, Protsenko S, Semiglazova T, Odintsova S, Zukov R, Lazarev S, Makarova Y, Nechaeva M, Sakaeva D, Andreev A, Tarasova A, Fadeyeva N, Shustova M, Kuryshev I. Novel PD-1 inhibitor prolgolimab: expanding non-resectable/metastatic melanoma therapy choice. Eur J Cancer. 2021 May;149:222-232. doi: 10.1016/j.ejca.2021.02.030. Epub 2021 Apr 17. PMID 33872982